CLINICAL TRIAL: NCT03445247
Title: An Investigation on the Effects of Extracorporeal Low-intensity Shockwave Therapy on Protenuria, Renal Function, and Blood Pressure in Type 2 Diabetic Patients in Stage 3-4 Chronic Kidney Disease
Brief Title: Extracorporeal Low-intensity Shockwave in Diabetic Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104-7771A
Record Dates: First submitted 2018-01-29; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2017-07

CONDITIONS: Diabetic Nephropathy Type 2
Keywords: Diabetic Nephropathies; Extracorporeal low intensity shockwave therapy; Proteinuria
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): No intervention, no placebo, but do the same blood tests and examinations as experiment group at the same time points
  Interventions: Other: Extracorporeal low-intensity shockwave
- Extracorporeal low-intensity shockwave group (Experimental): with 12 times extracorporeal low intensity shockwave therapy and do the blood test and assessments at baseline, 3, 6, 12 m after initiation of therapy.
  Interventions: Other: Extracorporeal low-intensity shockwave

INTERVENTIONS:
Other: Extracorporeal low-intensity shockwave — Omnispec device to give a total of 1200 shockwaves, with low energy density at 0.1 mj/mm2 and a frequency of 120 shocks/min per kidney per treatment session, totally 12 times.

SUMMARY:
In the current study, we use extracorporeal low-intensity shockwave therapy (ESWT) to treat on patients with type 2 diabetes in stage 3-4 chronic kidney disease and see whether it can improve the proteinuria, renal function, and blood pressure compared to baseline and control group.

DETAILED DESCRIPTION:
Diabetic nephropathy is the major contributor to end stage renal disease worldwide. Extracorporeal shock wave treatments (ESWT) with low-intensity was reported to be beneficial in inducing cell regeneration and reducing inflammation and have been successfully used for bone fracture, cardiac ischemia, and erectile disorders. In this study, sixty patients with stage III & IV (15<=estimated glomerular filtration rate (eGFR)<60 ml/min/1.73m2) will be recruited and allocated to control and experimental groups in a 1:1 ratio. In experiment group, a total of 1200 shockwaves, with low energy density 0.1mj/mm2 and a frequency of 120 shocks/min, will be applied per kidney per treatment session. The treatment will be given twice a week for 3 consecutive weeks, followed by 3 weeks of recess and an additional series of 6 sessions (totally 12 times). Patients in each group will be evaluated with eGFR, urine protein-creatinine ration, blood pressure, and biochemistry data at the beginning (index day) and 12 months after starting of the therapy. (Outcome time point: 12 months)

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 y/o or <80 y/o
2. Diagnosed as type 2 diabetes.
3. Baseline HbA1C <7.5%
4. Baseline glomerular filtration rate (eGFR) ≧15 and <60 ml/min/1.73m2
5. Baseline urine albumin-to-creatinine ratio (UACR) >30 and <3000 mg/g
6. Subject receives ACEi or ARB for 3 months before enrollment
7. Subject is willing to sign the permit and receive 12 times shockwave therapy

Exclusion Criteria:

1. Subject is pregnant or breast feeding
2. Subject has cancer or chronic inflammatory disease
3. Subject has bleeding tendency, eg thrombocytopenia, PT INR > 2.5
4. Subject has active urinary tract infection or other active infections
5. Subject's sBP>160mmHg or dBP>100mmHg
6. Subject has stroke, cardiac infection or arrhythmia in 6 months before enrollment
7. Subject has local inflammation or infection over treatment areas
8. Subject has pacemaker or other metal implants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
changes of estimated glomerular filtration rate | 12 month
  using Modification of Diet in Renal Disease (MDRD) equation, which is eGFR (mL/min/1.73m2) = 175 × serum creatinine-1.154 × age-0.203× 0.742 (if female) to evaluate renal function
changes of proteinuria | 12 month
  using spot urine albumin- and protein-creatinine ratio

SECONDARY OUTCOMES:
changes of systolic and diastolic blood pressure | 12 month
  Let patients rest for 15 mins and check blood pressure using same sphygmomanometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang-Gung Memorial Hospital, Kaohsiung City, Please Select, Taiwan

REFERENCES:
- [Derived] Klomjit N, Lerman A, Lerman LO. It Comes As a Shock: Kidney Repair Using Shockwave Therapy. Hypertension. 2020 Dec;76(6):1696-1703. doi: 10.1161/HYPERTENSIONAHA.120.14595. Epub 2020 Nov 2. PMID 33131308